CLINICAL TRIAL: NCT06345781
Title: Abdominal Functional Electrical Stimulation to Improve Bowel Function in Spinal Cord Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Craig Hospital (Other)
Collaborators: Neuroscience Research Australia (Other)
Responsible Party: Principal Investigator, Candace Tefertiller, Executive Director of Research and Evaluation, Craig Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2174433-1
Record Dates: First submitted 2024-03-28; First posted 2024-04-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Spinal Cord Injuries; Neurogenic Bowel
Keywords: Spinal Cord Injury; Functional Electrical Stimulation (FES); Neurogenic Bowel
MeSH Terms: conditions — Spinal Cord Injuries; Neurogenic Bowel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Abdominal Functional Electrical Stimulation (Experimental): All participants enrolled will receive the intervention.
  Interventions: Behavioral: Abdominal Functional Electrical Stimulation

INTERVENTIONS:
Behavioral: Abdominal Functional Electrical Stimulation — Functional electrical stimulation electrodes will be applied to the abdomen during a bowel program to assess effects of stimulation on bowel management time.

SUMMARY:
The primary objective of this study is to gather information about the effectiveness of abdominal FES to improve bowel management time (BMT) for people with chronic SCI. This study will also evaluate whether abdominal FES can improve: 1) bowel-related quality of life, 2) participant-reported bowel function, 3) bowel management strategy, 4) bladder symptoms, and 5) unplanned hospital admissions. In addition, we will also explore participant perspectives and experiences about the stimulation sessions and use of the device.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic SCI (> 12 months since injury) above the level of T11
2. > 18 years of age
3. a measurable and consistent start and end event is determinable for the bowel routine

   * Start events include: 1) enema insertion, 2) digital stimulation, 3) hot drink or initiation of the gastrocolic reflex, 3) abdominal massage, or 4) other, as determined by the participant and research team.
   * Ending events include: 1) final digital stimulation, 2) when evacuation has ceased, or 3) other, as determined by the participant and research team.
4. Portable smart device with video capabilities and internet access
5. Willingness to access and/or download Zoom (videoconferencing software)

Exclusion Criteria:

1. American Spinal Injuries Association (ASIA) Impairment Scale (AIS) E
2. Self-reported bowel management time (BMT) of <30 minutes
3. Current bowel conditions such as gastro-esophageal reflux, bowel obstruction, Crohn's disease, or diverticulitis
4. Physical obstacles that prevent AFES (e.g., pregnancy, abdominal trauma, cardiac pacemaker, or other implanted electromedical devices)
5. Stoma or colostomy
6. No response to AFES (e.g., lower motor neuron impairment)
7. History of gastrointestinal surgery within the past 3 months
8. Severely obese participants (>40 BMI)
9. Primary language other than English
10. Previous history of uncontrolled, recurrent episodes of AD
11. Resting systolic blood pressure (BP) reported as >140 mmHg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-04-30 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Bowel Management Time (BMT) | Daily (Weeks 1-10)
  This is measured by recording start and end time of bowel management session in study diary.

SECONDARY OUTCOMES:
Bowel Management Strategy | Daily (Weeks 1-10)
  This will be measured via analysis of daily diary entries regarding bowel movements (time taken and frequency), dietary changes or inconsistencies, and use of laxatives and manual procedures. The bowel diary will be completed daily throughout the study by participants and/or their caregivers.
Stimulation Dose | During active stimulation period (Weeks 3-7)
  This will be recorded by the participant. Participants will be asked to record the total time of active stimulation as displayed by the stimulation counter/timer and the intensity of the stimulation (milliamps) for each BM session in their bowel diary. The stimulation device will also record number of times the device button is depressed and duration in seconds, which can be downloaded at a later date by the research team providing further detail on stimulation dose.
EuroQoL 5 Dimension 5 Level (EQ-5D-5L) Questionnaire | Week 1, Week 3, Week 7, Week 10
  Quality of Life measure
International Spinal Cord Society's (ISCoS) International SCI Bowel Function Basic Data Set Questionnaire | Week 1, Week 3, Week 7, Week 10
  This instrument measures participant-reported bowel function bowel function.
Visual Analog Scale (VAS) | Week 1, Week 3, Week 7, Week 10
  This instrument measures participant perceptions of bowel function satisfaction on a rating scale from 0-100.
Neurogenic Bladder Symptom Score (NBSS) | Week 1, Week 3, Week 7, Week 10
  This instrument measures neurogenic bladder symptoms
Intervention Acceptability | Week 7
  Qualitative and quantitative analysis of abdominal functional stimulation (AFES) use will be measured at the end of the active trial period, using both open-ended and 10-scored theoretical framework of acceptability questions to gain the perspective of people with lived experience of SCI on the use of AFES during a bowel routine
Intervention Safety | Daily (Weeks 0-10)
  This will be determined by the reporting and summarization of any adverse events associated with the interventions. Participants will be instructed to record any adverse events in their bowel diaries and to call study staff immediately to review. Unplanned hospital visits will also be recorded in the study diary.

CONTACTS AND LOCATIONS:
Locations (1):
- Craig Hospital, Englewood, Colorado, United States

IPD SHARING:
Plan to Share IPD: No